CLINICAL TRIAL: NCT00388973
Title: A Multi-Centre, Double-Blind, Randomised, Parallel-Group, Placebo-Controlled Phase III Study of the Efficacy and Safety of Quetiapine Fumarate Sustained Release (Seroquel SR) in the Treatment of Elderly Patients With Major Depressive Disorder
Brief Title: Efficacy and Safety Study of Seroquel SR in the Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Martin Brecher, Seroquel Medical Science Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1448C00014; EUDRACT No: 2006-001196-38
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Results first posted 2010-04-01 (Estimated); Last update posted 2010-04-01 (Estimated); Status verified 2010-03

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine

SUMMARY:
The primary purpose of this study is to evaluate whether treatment with (SEROQUEL SR) quetiapine fumarate sustained release (SR) for 9 weeks compared to placebo will improve depressive symptoms in elderly patients with major depressive disorder.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 66 years or older, with a documented clinical diagnosis of MDD.

Exclusion Criteria:

* The presence of dementia or mental disorder other than MDD within 6 months of enrolment,
* Uncontrolled hypertension, substance or alcohol abuse
* A current diagnosis of cancer or a current or past diagnosis of stroke

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 338 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Datto, MD, Study Director — AstraZeneca
Locations (43):
- United States (13):
  - Research Site, Birmingham, Alabama
  - Research Site, San Diego, California
  - Research Site, Fort Myers, Florida
  - Research Site, Gainsville, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Roswell, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, Brooklyn, New York
  - Research Site, Eugene, Oregon
  - Research Site, Jenkintown, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, San Antonio, Texas
- Argentina (6):
  - Research Site, City Bell, Buenos Aires
  - Research Site, La Plata, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Mendoza, Mendoza Province
  - Research Site, Buenos Aires
  - Research Site, Capital Federal
- Estonia (3):
  - Research Site, Tartu, Estonia
  - Research Site, Tallinn
  - Research Site, Viljandi
- Finland (6):
  - Research Site, Helsinki, Finland
  - Research Site, Tampere, Finland
  - Research Site, Jarvenpaa
  - Research Site, Kuopio
  - Research Site, Salo
  - Research Site, Seinäjoki
- Russia (8):
  - Research Site, Arkhangelsk
  - Research Site, Izhevsk
  - Research Site, Lipetsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Stavropol
- Ukraine (7):
  - Research Site, Hlevakha, Kyiv Oblast
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kiev
  - Research Site, Luhansk
  - Research Site, Odesa
  - Research Site, Vinnitsa

REFERENCES:
- [Derived] Weisler R, Montgomery SA, Earley WR, Szamosi J, Eriksson H. Extended release quetiapine fumarate in patients with major depressive disorder: suicidality data from acute and maintenance studies. J Clin Psychiatry. 2014 May;75(5):520-7. doi: 10.4088/JCP.13m08624. PMID 24816198
- [Derived] Weisler R, McIntyre RS. The role of extended-release quetiapine fumarate monotherapy in the treatment of patients with major depressive disorder. Expert Rev Neurother. 2013 Nov;13(11):1161-82. doi: 10.1586/14737175.2013.846520. PMID 24175720
- [Derived] Montgomery SA, Altamura AC, Katila H, Datto C, Szamosi J, Eriksson H. Efficacy of extended release quetiapine fumarate monotherapy in elderly patients with major depressive disorder: secondary analyses in subgroups of patients according to baseline anxiety, sleep disturbance, and pain levels. Int Clin Psychopharmacol. 2014 Mar;29(2):93-105. doi: 10.1097/YIC.0000000000000007. PMID 24162081
- [Derived] Locklear JC, Svedsater H, Datto C, Endicott J. Effects of once-daily extended release quetiapine fumarate (quetiapine XR) on quality of life and sleep in elderly patients with major depressive disorder. J Affect Disord. 2013 Jul;149(1-3):189-95. doi: 10.1016/j.jad.2013.01.021. Epub 2013 Apr 29. PMID 23639212
- [Derived] Katila H, Mezhebovsky I, Mulroy A, Berggren L, Eriksson H, Earley W, Datto C. Randomized, double-blind study of the efficacy and tolerability of extended release quetiapine fumarate (quetiapine XR) monotherapy in elderly patients with major depressive disorder. Am J Geriatr Psychiatry. 2013 Aug;21(8):769-84. doi: 10.1016/j.jagp.2013.01.010. Epub 2013 Feb 6. PMID 23567397

RESULTS

PARTICIPANT FLOW:
Recruitment Details: International multi-center study, 53 sites recruited between Sept 2006 and Dec 2007
Pre-assignment Details: Screening for eligibility and wash-out of restricted medications. At least moderate depression symptoms assessed by the Hamilton Rating Scale for Depression
Groups:
- Quetiapine XR: Quetiapine fumarate XR - flexibly dosed (50 - 300 mg)
- Placebo: Placebo
Period: Overall Study
Arm/Group | Quetiapine XR | Placebo
Started | 166 (Randomized) | 172 (Randomized)
Completed Study | 110 | 114
Completed | 110 (Completed 9-week treatment and 2 week follow-up) | 114 (Completed 9-week treatment and 2 week follow-up)
Not Completed | 56 | 58
Not completed — Adverse Event | 16 | 6
Not completed — Lack of Efficacy | 1 | 12
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 14 | 17
Not completed — Study specific Discontinuation Criteria | 0 | 1
Not completed — Did not complete 61 days of treatment | 5 | 4
Not completed — Left region | 0 | 1
Not completed — Did not complete 2-week follow-up visit | 17 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine XR | Placebo | Total
Number analyzed (Participants) | 166 | 172 | 338
Age, Customized [Number; unit: Participants]
  66 to 75 years | 135 | 137 | 272
  >75 years | 31 | 35 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 120 | 236
  Male | 50 | 52 | 102
Region of Enrollment [Number; unit: Participants]
  Europe | 124 | 126 | 250
  North America | 24 | 27 | 51
  South America | 18 | 19 | 37
DSM IV diagnosis [Number; unit: Participants]
  296.2x - Major depressive disorder, single episode | 27 | 25 | 52
  296.3x - Major depressive disorder, recurrent | 139 | 147 | 286

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score to Week 9.
Description: MADRS total score (0-60 units), where lower scores indicate less depressive symptoms, calculated as Week 9 value - baseline value.
Time Frame: Baseline to Week 9
Population: All randomized patients who took at least one dose of study medication and had at least one post baseline assessment, with last observation carried forward to week 9 for patients who did not complete the study.
Measure: Least Squares Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 164 | 171
units on scale | -16 (8) | -9 (8)

2. Secondary Outcome: Change From Baseline in Health-related Quality of Life, Enjoyment and Satisfaction (Q-LES-Q)
Description: Q-LES-Q as percent of maximum (0 to 100%) calculated as Week 9 - baseline, where higher values indicate better quality of life.
Time Frame: Baseline to Week 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Percentage of Improvement
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 164 | 171
Percentage of Improvement | 17 (14) | 9 (14)

3. Secondary Outcome: Change From Baseline for Satisfaction With Medication From Quality of Life, Enjoyment, Satisfaction Questionaire (Q-LES-Q)
Description: Item 15 the Quality of Life, Enjoyment Satisfaction Questionnaire (score 1 least -5 best) on Q-LES-Q, calculated as Week 9 value - baseline value
Time Frame: Baseline to Week 9
Population: All randomized patients who took at least one dose of study medication and had at least one post baseline assessment, with last observation carried forward to week 9 for patients who did not complete the study. Patients not on medication at baseline would have left the item blank and therefore no change from baseline could be calculated
Measure: Median (Full Range); unit: units on scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 55 | 70
units on scale | 0 [-1 to 2] | 0 [-3 to 3]

4. Secondary Outcome: Change From Baseline in Anxiety Symptoms Measured by Hamilton Anxiety 14 Item Scale (HAM-A)
Description: Change in HAM-A total score (total score 0-56), calculated as Week 9 value - baseline value, where lower scores indicate less anxiety.
Time Frame: Baseline to Week 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 164 | 171
units on a scale | -11 (6) | -5 (8)

5. Secondary Outcome: Change From Baseline in Sleep Quality as Measured by the Pittsburgh Sleep Quality Index
Description: The Pittsburgh Sleep Quality Index is an eighteen questionnaire scored with 7 sleep component scores each on a 0 to 3 scale, total score range from 0 to 21, worst value 21, best value 0
Time Frame: Baseline to Week 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 164 | 171
units on scale | -6 (4) | -3 (4)

6. Secondary Outcome: Change From Baseline in Suicidal Thoughts as Measured by Montgomery-Asberg Depression Rating Scale (MADRS) Item 10
Description: The suicide item is a single item of the Montgomery-Asberg Depression Rating Scale with a range of values from 0 to 6, worst value 6, best value 0
Time Frame: Baseline to Week 9
Population: as for outcome 1
Measure: Median (Full Range); unit: units on scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 164 | 171
units on scale | 0 [-2 to 2] | 0 [-2 to 5]

7. Secondary Outcome: Change From Baseline in Somatic Symptoms Cluster From the Hamilton Anxiety Scale (HAM-A)
Description: The Somatic symptom Cluster of the Hamilton Anxiety Scale is a 7 item cluster associated with somatic symptoms *somatic muscular, somatic sensory, cardiovascular system, respiratory system, gastrointestinal system, genitourinary system, autonomic system) with a range of values from 0 to 28, worst value 28, best value 0
Time Frame: Baseline to Week 9
Population: as for outcome 1
Measure: Median (Full Range); unit: units on scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 164 | 171
units on scale | -4 (-15.7) [-15 to 7] | -2 (-14.6) [-14 to 6]

8. Secondary Outcome: Tolerability as Measured by Adverse Event Withdrawals During Treatment
Time Frame: Baseline to Week 9
Population: All Randomized patients.
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 166 | 172
Participants | 16 | 7

ADVERSE EVENTS:
Arm/Group | Quetiapine XR | Placebo
Serious Adverse Events (participants affected / at risk) | 4/166 | 2/172
Other Adverse Events (participants affected / at risk) | 133/166 | 54/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine XR (N=166) | Placebo (N=172)
Depression (Psychiatric disorders) | 0 | 2
Depressive Symptom (Psychiatric disorders) | 1 | 0
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine XR (N=166) | Placebo (N=172)
Dizziness (Nervous system disorders) | 32 | 26
Dry Mouth (Gastrointestinal disorders) | 34 | 0
Headache (Nervous system disorders) | 35 | 28
Somnolence (Nervous system disorders) | 55 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees to collaborate in good faith with AstraZeneca with regard to the contents and formation of any publication or disclosure to be made by the PI and to pay due consideration to the comments, views and opinions offered by AstraZeneca.